CLINICAL TRIAL: NCT06857669
Title: Breast Cancer Diagnosis Using Optical Techniques
Brief Title: Clinical Explorative Optical Breast Investigations
Acronym: CLEO-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other); Unilabs (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Dnr 2019-04840
Record Dates: First submitted 2025-01-07; First posted 2025-03-04 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Benign Breast Tumors; Malignant Breast Tumours; Healthy
Keywords: breast; optical imaging; photoacoustic; spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Diffuse reflectance spectroscopy or Photoacoustic imaging) (Experimental): In part I, 30 breast specimens will be examined by DRS (ex-vivo). In part II, 30 breast specimens will be examined by both DRS and PAI (ex-vivo). In part III, 30 individuals will be examined by PAI (in-vivo).
  Interventions: Diagnostic Test: Diffuse reflectance spectroscopy and Photoacoustic imaging,

INTERVENTIONS:
Diagnostic Test: Diffuse reflectance spectroscopy and Photoacoustic imaging, — The photoacoustic imaging/diffuse reflectance spectroscopy techniques used in this study have a broader wavelength spectrum. The photoacoustic set-up can generate an optical and an ultrasound image simultaneously.

SUMMARY:
This study evaluates diffuse reflectance spectroscopy and photoacoustic imaging for differentiating healthy, benign, and malignant breast tissue by identifying their optical profiles.

DETAILED DESCRIPTION:
Breast cancer is the most prevalent cancers among women worldwide. Current diagnostic modalities have notable limitations. Mammography exposes patients to harmful ionising radiation whilst MRI often requires intravenous contrast agents. Additionally, diagnosing breast cancer frequently relies on invasive biopsies, which can cause patient discomfort.

This study investigates the potential use of two optical modalities, diffuse reflectance spectroscopy (DRS) and photoacoustic imaging (PAI), as non-invasive diagnostic tools for breast tissue analysis. Advantages include use of non-ionising radiation, contrast-free imaging, and the ability to assess tissue properties in detail.

DRS is a non-image based hand-held modality that utilises white light to generate optical signals. PAI is a hybrid biomedical imaging modality that combines traditional ultrasound with optical imaging. The latter generates a functional image that can potentially assess oxygenation levels which is known to be different in healthy vs cancerous tissue.

The study will focus on analysing three types of human breast tissues: healthy tissue, benign lesions (such as fibroadenomas), and malignant lesions (invasive breast carcinomas). By identifying the unique optical signatures of each tissue type, the research aims to evaluate the feasibility of these optical techniques as complementary tool to traditional imaging methods for diagnosing or monitoring breast cancer in the future.

ELIGIBILITY:
Inclusion Criteria:

* solitary malignant or benign biopsy verified tumour > 1 cm
* understands written and oral Swedish

Exclusion Criteria:

* previous breast surgery
* has received neoadjuvant chemotherapy
* skin burns in on the chest

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of study subjects with correctly classified breast tissue type with PAI/DRS | 30 days
  To evaluate if optical techniques (DRS/PAI) can differentiate between three breast tissue types, namely healthy, benign and malignant tissue. Differences in the optical tissue-properties will be compared to histopathological evaluation.

SECONDARY OUTCOMES:
Optical signal in relation to photoacoustic imaging depth | 2 days
  Signal intensity will be measured at 5 mm intervals; from skin surface to a depth of approximately 35 mm.
To assess oxygenation levels across three breast tissue types using PAI | Immediately after photoacoustic imaging acquisition
  The percentage of oxygenation within a region of interest (ROI)

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Zackrisson, MD, PhD, Principal Investigator — Region Skane, Lund University
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
The data used in this study contains sensitive information about the study participants and they did not provide consent for public data sharing. A minimal data set could, however, be shared by request from a qualified academic investigator for the sole purpose of replicating the present study, provided the data transfer is in agreement with EU legislation on the general data protection regulation and approval by the Swedish Ethical Review Authority.

REFERENCES:
- [Result] Chaudhry N, Albinsson J, Cinthio M, Kroll S, Malmsjo M, Ryden L, Sheikh R, Reistad N, Zackrisson S. Breast Cancer Diagnosis Using Extended-Wavelength-Diffuse Reflectance Spectroscopy (EW-DRS)-Proof of Concept in Ex Vivo Breast Specimens Using Machine Learning. Diagnostics (Basel). 2023 Sep 28;13(19):3076. doi: 10.3390/diagnostics13193076. PMID 37835819
- See also: photoacoustic center at Lund University — https://www.photoacoustics.lu.se/lund-university-photoacoustic-center